CLINICAL TRIAL: NCT02640950
Title: An Open Label Trial of TMS Therapy for Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Scott T. Aaronson, M.D, Director, Clinical Research Programs, Sheppard Pratt Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 794736-5
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Results first posted 2022-05-12 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label TMS (Experimental): Active Transcranial Magnetic Stimulation
  Interventions: Device: NeuroStar TMS

INTERVENTIONS:
Device: NeuroStar TMS — Transcranial Magnetic Stimulation
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
Transcranial Magnetic Stimulation (TMS) is an increasingly accepted neurostimulation- based treatment for major depressive disorder. While there is a growing anecdotal database supporting its use in bipolar depression the investigators propose to collect open label efficacy and safety data in a small population of patients with clinically verified bipolar disorder.

DETAILED DESCRIPTION:
The investigators propose to screen patients with bipolar depression I or II, who are already on acceptable mood stabilization. They may or may not be on antidepressants at the time of screening but subjects on antidepressants would be taken off them before completing the screening phase. Those patients who have a depression of at least moderate severity without significant symptoms of activation or mania will be started on a course of open label TMS treatment of up to 35 sessions. Safety and efficacy assessments will be done weekly. Patients will complete a course of treatment when they meet remission criteria (MADRS score < 10) or at the end of 30 treatments, whichever comes first. Patient who are still judged to be improving between treatment 25 and treatment 30 will be eligible to complete up to five addition treatments as the discretion of each site's principal investigator. Patients who meet response criteria (MADRS score decreases by at least 50%) will complete the full course of 30 to 35 TMS sessions. Patients will be withdrawn for safety concerns, particularly the onset of activation suggestive of mania or a mixed state.

Patients who meet response or remission criteria will be followed monthly for up to six months to evaluate the durability of response. They will be on standard mood stabilizing medications and psychotherapy per their clinician's discretion.

ELIGIBILITY:
Inclusion Criteria- Phase II:

1. Must be at least 18 years old.
2. Must meet DSM-5 criteria for bipolar (either I or II) depression by clinical interview and M.I.N.I. The duration of the current depressive episode must be at least 4 weeks and no longer than 3 years in length.
3. Should have a MADRS score of at least 20 at screening, an YMRS score of less than 12 and a CGI score of at least 4.
4. Must have signed the informed consent document and have a level of understanding sufficient to provide informed consent and to communicate with the investigator and site personnel.
5. Must be on a mood stabilizer acceptable to the study physician which is consistent with their diagnosis. The mood stabilizer must be at a stable dose for at least four days before starting TMS treatment.
6. If female of childbearing potential, patients must

   1. have a negative urine pregnancy test at screening, and
   2. not be nursing or planning a pregnancy, and
   3. be on a medically acceptable method of birth control acceptable to the principal investigator.

Choices of contraception that meet the study requirements are

* Intrauterine device
* Hormonal contraception (estrogen-containing birth control pills, Vaginal ring, patch, injections or implants)
* Latex condom with spermicide
* Diaphragm with spermicide
* Cervical cap with spermicide

Females of childbearing potential who are abstinent can enroll in the study.

Exclusion Criteria- Phase II:

1. May not be directly affiliated with Sheppard Pratt Clinical Research Programs or be immediate family of Research Programs personnel.
2. Must not have another primary Axis I diagnosis.
3. The subject must not have stopped an antidepressant less than two weeks before starting TMS treatment or unable to discontinue antidepressant therapy.
4. Should have no previous history of psychosis or substance dependence or abuse within the six months prior to Screening
5. Presence of an Axis II disorder felt by the investigator to potentially interfere with study compliance would exclude a potential participant.
6. Should not have prior intolerance of TMS or significant lack of response to adequate trials of TMS.
7. Should not have a lifetime history of lack of response to ECT or VNS.
8. Should not have any medical condition likely to interfere with safe study participation.
9. Women of child-bearing potential who are not using a medically accepted means of contraception when engaging in sexual intercourse are excluded, as well as women who are pregnant or breast-feeding.
10. Positive urine screen for any substance of abuse will exclude a patient, with the exception of benzodiazepines. A satisfactory explanation in the opinion of the investigator along with a negative repeat screen prior to Visit 2 is possibly acceptable.
11. Current suicide risk, as evidenced:

    1. It is the judgment of the investigator that the patient may be at risk for suicide
    2. The patient has rated a "yes" to question 4 or question 5 on the Screening C-SSRS
    3. The patient has attempted suicide within the past 12 months prior to Screening.
12. History of head injury, epilepsy or seizure disorder, non-removable metallic implants or objects in or around the head.

Inclusion Criteria- Phase III Patients who meet MADRS criteria for response or remission will enter Phase III, the six month follow-up phase of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-12; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Aaronson, MD, Principal Investigator — Sheppard Pratt Health System
Locations (2):
- United States (2):
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Department of Psychiatry and Psychology, Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aaronson ST, Goldwaser EL, Croarkin PE, Geske JR, LeMahieu A, Sklar JH, Kung S. A Pilot Study of High-Frequency Transcranial Magnetic Stimulation for Bipolar Depression. J Clin Psychiatry. 2024 May 20;85(2):23m15056. doi: 10.4088/JCP.23m15056. PMID 38780536

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Bipolar (I or II) Depression: Adults with bipolar (I or II) depression, per DSM-5 criteria, were recruited at Sheppard Pratt and Mayo Clinic between December 2015-February 2020 for TMS. Standardized treatment protocols employed 6 weeks of 10 Hz TMS to the left dorsolateral prefrontal cortex at 120% of motor threshold with 3,000 pulses per session in 4 second trains with intertrain intervals of 26 seconds. All patients were treated concurrently with a mood stabilizer. The primary outcome measure was the Montgomery-Asberg Depression Rating Scale (MADRS). Response and remission were defined as MADRS score reductions of ≥ 50% or score ≤10, respectively. We examined response, remission, and potential contributing factors with multivariate and logistic regression models.
Period: Overall Study
Arm/Group | Patients With Bipolar (I or II) Depression
Started | 31
Completed | 29
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Bipolar (I or II) Depression
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31
Montgomery-Åsberg Depression Rating Scale [Number; unit: Number of participants] — The MADRS is a clinician rated scale measuring depression severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60; higher scores denote greater severity. A decrease in MADRS score of at lease 50% will be considered a response to treatment. A MADRS score of less than 10 will be considered remission.
  Number of participants
    Participants in remission at baseline | 0
    Participants responding at baseline | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Who Respond or Remit After 30 to 35 Treatments Based Off of the Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: The MADRS is a clinician rated scale measuring depression severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60; higher scores denote greater severity. A decrease in MADRS score of at lease 50% will be considered a response to treatment. A MADRS score of less than 10 will be considered remission.
Time Frame: Up to 7 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Bipolar (I or II) Depression: Adults with bipolar (I or II) depression, per DSM-5 criteria, were recruited at Sheppard Pratt and Mayo Clinic between December 2015 -February 2020 for TMS. Standardized treatment protocols employed 6 weeks of 10 Hz TMS to the left dorsolateral prefrontal cortex at 120% of motor threshold with 3,000 pulses per session in 4 second trains with intertrain intervals of 26 seconds. All patients were treated concurrently with a mood stabilizer. The primary outcome measure was the Montgomery-Asberg Depression Rating Scale (MADRS). Response and remission were defined as MADRS score reductions of ≥ 50% or score ≤10, respectively. We examined response, remission, and potential contributing factors with multivariate and logistic regression models.
Arm/Group | Patients With Bipolar (I or II) Depression
Number analyzed (Participants) | 31
Participants
  Response Criteria: Number meeting criteria | 27
  Response Criteria: Number of non-responders | 4
  Remission Criteria: Number meeting criteria | 23
  Remission Criteria: Number of non-responders | 8
Statistical Analysis 1: Comparison: Patients With Bipolar (I or II) Depression; Paired t-test of pre and post treatment scores on MADRS; Test type: Superiority; p < 0.001, t-test, 2 sided — Paired t test for pre and post treatment scores for all subjects

2. Primary Outcome: The Percentage of Patients Who Meet Criteria for Onset of Manic Symptoms Based on the Young Mania Rating Scale (YMRS).
Description: The Young Mania Rating Scale (YMRS) is used to determine the severity of a patient's mania. The score for the YMRS ranges form 0 to 60. Scores of 13-19 indicate minimal manic symptoms, 20-25 is mild mania, 26-37 is moderate mania, and 38-60 is severe mania. A YMRS score of 14 or greater will be used for criteria of onset of manic symptoms. The patients will be separated based on their diagnostic category of either Bipolar I Disorder or Bipolar II Disorder.
Time Frame: Up to 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Bipolar (I or II) Depression
Number analyzed (Participants) | 31
Participants
  Bipolar I Disorder | 20
  Bipolar II Disorder | 11
  Bipolar I Participants with Onset of Maniac Symptoms | 0
  Bipolar II Participants with Onset of Maniac Symptoms | 0
Statistical Analysis 1: Comparison: Patients With Bipolar (I or II) Depression; Test type: Other — Descriptive Frequencies Analysis; A frequencies analysis was conducted to determine the number of participants that were diagnosed with BP I and BP II as well as the number of participants that developed an onset of maniac symptoms during the 7 week treatment period

3. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) to Calculate Percentage of Patients Meeting Response Criteria
Description: The Hamilton Depression (HAM-D) Rating Scale is a scale used to measure one's depression. The scoring from the scale ranges 0 to 53. Higher scores indicate that a person is more depressed. The scoring ranges from 0-7 is normal, 8-13 is mild depression, 14-18 is moderate depression, 19-22 severe depression, and greater than or equal to 23 is very severe depression. The HAM-D response criteria will be based off a HAM-D score drop of at least 50%. Remission HAM-D score will be 7 or less.
Time Frame: Up to 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Bipolar (I or II) Depression
Number analyzed (Participants) | 31
Participants
  Remission : Met criteria | 21
  Remission : Non-responders | 10
  Response : Met criteria | 24
  Response : Non-responders | 7

4. Secondary Outcome: Clinical Global Impression (CGI) to Calculate Percentage of Patients Meeting Response Criteria
Description: The Clinical Global Impression (CGI) Scale is used to determine the severity of a patient's depression. The scoring for the scale ranges from 1 to 7, where 1 indicates that the patient is normal and 7 indicates a severe depression.
  Remission criteria for the CGI score will be a 2 or less.
  Responders and remitters will also be followed for six months after the final treatment to see the durability of response. Percentage of patients' meeting relapse criteria will be calculated.
Time Frame: Up to 7 weeks and 6 Month Follow Up
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Bipolar (I or II) Depression
Number analyzed (Participants) | 31
Participants
  Remission Criteria During 7 Week Treatment: Met criteria | 27
  Remission Criteria During 7 Week Treatment: Did not meet criteria | 4
  Relapse Criteria During 6 Month Follow Up: Met criteria | 9
  Relapse Criteria During 6 Month Follow Up: Did not meet criteria | 22

5. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) to Average Number of Treatments Needed to Meet Remission
Description: For the patients meeting remission criteria (Total Number = 21) , we will calculate the number of treatments required to achieve remission. Patients who only meet response criteria will be treated for 30 to 35 sessions.
Time Frame: 7 Weeks
Measure: Mean (Standard Deviation); unit: Number of Treatments
Arm/Group | Patients With Bipolar (I or II) Depression
Number analyzed (Participants) | 21
Number of Treatments | 25.76 (5.02)

6. Secondary Outcome: Clinical Global Impression (CGI) to Calculate Average Number of Treatments Needed to Meet Remission
Description: For the patients meeting remission criteria (Total Number = 27) , we will calculate the number of treatments required to achieve remission. Patients who only meet response criteria will be treated for 30 to 35 sessions.
Time Frame: 7 Weeks
Measure: Mean (Standard Deviation); unit: Number of Treatments
Arm/Group | Patients With Bipolar (I or II) Depression
Number analyzed (Participants) | 27
Number of Treatments | 26.48 (4.45)

ADVERSE EVENTS:
Time Frame: Six months
Groups:
- Patients With Bipolar (I or II) Depression: Thirty-one adults (13M/18F; age: 42.2[14.3]) with bipolar (I or II) depression, per DSM-5 criteria, were recruited at Sheppard Pratt and Mayo Clinic between December 2015-February 2020 for TMS. Standardized treatment protocols employed 6 weeks of 10 Hz TMS to the left dorsolateral prefrontal cortex at 120% of motor threshold with 3,000 pulses per session in 4 second trains with intertrain intervals of 26 seconds. All patients were treated concurrently with a mood stabilizer. The primary outcome measure was the Montgomery-Asberg Depression Rating Scale (MADRS). Response and remission were defined as MADRS score reductions of ≥ 50% or score ≤10, respectively. We examined response, remission, and potential contributing factors with multivariate and logistic regression models.
Arm/Group | Patients With Bipolar (I or II) Depression
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Bipolar (I or II) Depression (N=31)
Agitation (Psychiatric disorders) | 1 (1) — Agitation

LIMITATIONS AND CAVEATS:
Open label trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT02640950/Prot_SAP_000.pdf